CLINICAL TRIAL: NCT03117998
Title: A Randomized, Placebo-controlled, Double-blind Study to Evaluate the Efficacy, Safety, and Pharmacodynamics of Multiple Doses of REMD-477 in Subjects With Type 1 Diabetes Mellitus
Brief Title: Multiple Dose Study to Evaluate the Efficacy, Safety and Pharmacodynamics of REMD-477 in Subjects With Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: REMD Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R477-202
Record Dates: First submitted 2017-04-10; First posted 2017-04-18 (Actual); Results first posted 2023-05-25 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Type1 Diabetes Mellitus
MeSH Terms: interventions — volagidemab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 35 mg REMD-477 (Experimental): Administered as a repeated subcutaneous (SC) doses in subjects with Type 1 Diabetes
  Interventions: Biological: REMD-477
- 70 mg REMD-477 (Experimental): Administered as a repeated SC doses in subjects with Type 1 Diabetes
  Interventions: Biological: REMD-477
- Matching placebo (Placebo Comparator): Administered as a repeated SC doses in subjects with Type 1 Diabetes
  Interventions: Biological: Placebo Comparator

INTERVENTIONS:
Biological: REMD-477 — Administered as repeated SC doses in subjects with Type 1 Diabetes
  Arms: 35 mg REMD-477; 70 mg REMD-477
Biological: Placebo Comparator — Administered as a repeated SC doses in subjects with Type 1 Diabetes
  Arms: Matching placebo

SUMMARY:
This is a randomized, placebo-controlled, double-blind study to evaluate the efficacy, safety, and pharmacodynamics (PD) of multiple doses of REMD-477 in subjects who have Type 1 diabetes and are currently receiving insulin treatment. This study will determine whether REMD-477 can decrease daily insulin requirements and improve glycemic control after 12 weeks of treatment in subjects diagnosed with Type 1 diabetes with fasting C-peptide < 0.7 ng/mL at Screening.

The study will be conducted at multiple sites in the United States. Approximately 150 subjects with type 1 diabetes on stable doses of insulin will be randomized in a 1:1:1 fashion into one of three treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between the ages of 18 and 65 years old, inclusive, at the time of screening;
* Females of non-child bearing potential must be ≥1 year post-menopausal (confirmed by a serum follicle-stimulating hormone (FSH) levels ≥ 40 IU/mL) or documented as being surgically sterile. Females of child bearing potential must agree to use two methods of contraception;
* Male subjects must be willing to use clinically acceptable method of contraception during the entire study;
* Body mass index between 18.5 and 32 kg/m2, inclusive, at screening;
* Diagnosed with Type 1 diabetes, based on clinical history or as defined by the current American Diabetes Association (ADA) criteria;
* HbA1c > 7% and < 10 % at screening;
* Fasting C-peptide < 0.7 ng/mL;
* Treatment with a stable insulin regimen for at least 8 weeks before screening with multiple daily insulin (MDI) injections or continue subcutaneous insulin infusion (CSII)
* Willing to use continuous CGM system (e.g. DexCom) throughout the study;
* Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) ≤ 1.5x upper limit of normal (ULN) at screening;
* Able to provide written informed consent approved by an Institutional Review Board (IRB).

Exclusion Criteria:

* History or evidence of clinically-significant disorder or condition that, in the opinion of the Investigator, would pose a risk to subject safety or interfere with the study evaluation, procedures, or completion;
* Significant organ system dysfunction (e.g., clinically significant pulmonary or cardiovascular disease, anemia [Hemoglobin < 10.0 g/dL], known hemoglobinopathies, and renal dysfunction [eGFR < 60 ml/min]);
* Any severe symptomatic hypoglycemic event associated with a seizure or requiring help from other people or medical facility in the past 6 months;
* Myocardial infarction, unstable angina, revascularization procedure, or cerebrovascular accident ≤12 weeks before screening;
* History of New York Heart Association Functional Classification III-IV cardiac disease;
* Current or recent (within 1 month of screening) use of diabetes medications other than insulin - subjects on an SGLT2 inhibitor should be discontinue the SGLT2 inhibitor during the Screening Period, at least 2 weeks prior to the start of the Lead-in Period;
* Use of steroids and/or other prescribed or over-the-counter medications that are known to affect the outcome measures in this study or known to influence glucose metabolism;
* Smokes > 10 cigarettes/day, and/or is unwilling to abstain from smoking during admission periods;
* Known sensitivity to mammalian-derived drug preparations, recombinant protein-based drugs or to humanized or human antibodies;
* History of illicit drug use or alcohol abuse within the last 6 months or a positive drug urine test result at screening;
* History of pancreatitis, pancreatic neuroendocrine tumors or multiple endocrine neoplasia (MEN) or family history of MEN;
* History of pheochromocytoma, or family history of familial pheochromocytoma;
* Known or suspected susceptibility to infectious disease (e.g. taking immunosuppressive agents or has a documented inherited or acquired immunodeficiency);
* Known history of positive for human immunodeficiency virus (HIV) antibodies, hepatitis B surface antigen (HbsAg), or hepatitis C antibodies (HepC Ab);
* Participation in an investigational drug or device trial within 30 days of screening or within 5 times the half-life of the investigational agent in the other clinical study, if known, whichever period is longer;
* Blood donor or blood loss > 500 mL within 30 days of Day 1;
* Women who are pregnant or lactating/breastfeeding;
* Unable or unwilling to follow the study protocol or who are non-compliant with screening appointments or study visits;
* Any other condition(s) that might reduce the chance of obtaining study data, or that might cause safety concerns, or that might compromise the ability to give truly informed consent

Other inclusion and exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2017-09-19 (Actual); Primary Completion 2021-03-05 (Actual); Study Completion 2021-03-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - AMCR Institute, Escondido, California
  - Marin Endocrine Care & Research, Greenbrae, California
  - Altman Clinical and Translational Research Institute, San Diego, California
  - Diablo Clinical Research, Walnut Creek, California
  - University of Colorado, Denver/Barbara Davis Center for Diabetes, Aurora, Colorado
  - Atlanta Diabetes Assoicates, Atlanta, Georgia
  - Washington University School of Medicine, St Louis, Missouri
  - Texas Diabetes & Endocrinology, Austin, Texas
  - Dallas Diabetes Research Center, Dallas, Texas
  - Clinical Trials of Texas, San Antonio, Texas
  - Rainer Clinical Research Center, Renton, Washington

REFERENCES:
- [Derived] Santiago Padilla L, Schiattarella GG. Targeting HFpEF: Unlocking the Potential of Glucagon Receptor Blockade. Circ Res. 2024 Aug 16;135(5):629-631. doi: 10.1161/CIRCRESAHA.124.325130. Epub 2024 Aug 15. No abstract available. PMID 39146397

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A - 35 mg REMD-477; Part B - 35 mg REMD-477: Administered as a repeated subcutaneous (SC) doses in subjects with Type 1 Diabetes
  35 mg REMD-477: Administered as repeated SC doses in subjects with Type 1 Diabetes
- Part A - 70 mg REMD-477: Administered as a repeated SC doses in subjects with Type 1 Diabetes
  70 mg REMD-477: Administered as repeated SC doses in subjects with Type 1 Diabetes
- Part A - Matching Placebo: Administered as a repeated SC doses in subjects with Type 1 Diabetes
  Placebo Comparator: Administered as a repeated SC doses in subjects with Type 1 Diabetes
- Part B - 70 mg REMD-477: Administered as a repeated subcutaneous (SC) doses in subjects with Type 1 Diabetes
  70 mg REMD-477: Administered as repeated SC doses in subjects with Type 1 Diabetes
- Part B - Matching Placebo: Administered as a repeated subcutaneous (SC) doses in subjects with Type 1 Diabetes
  Placebo Comparator: Administered as a repeated SC doses in subjects with Type 1 Diabetes
Period: Overall Study
Arm/Group | Part A - 35 mg REMD-477 | Part A - 70 mg REMD-477 | Part A - Matching Placebo | Part B - 35 mg REMD-477 | Part B - 70 mg REMD-477 | Part B - Matching Placebo
Started | 25 | 25 | 25 | 26 | 26 | 27
Completed | 24 | 24 | 21 | 22 | 19 | 24
Not Completed | 1 | 1 | 4 | 4 | 7 | 3
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 3 | 3 | 0
Not completed — Physician Decision | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 4 | 0
Not completed — Subject noncompliance | 0 | 0 | 1 | 0 | 0 | 2
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A - 35 mg REMD-477 | Part A - 70 mg REMD-477 | Part A - Matching Placebo | Part B - 35 mg REMD-477 | Part B - 70 mg REMD-477 | Part B - Matching Placebo | Total
Number analyzed (Participants) | 25 | 25 | 25 | 26 | 26 | 27 | 154
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (13.1) | 43 (13.7) | 45 (14.8) | 42 (13.8) | 38 (14.1) | 42 (14.8) | 42 (14.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 14 | 15 | 15 | 17 | 12 | 92
  Male | 6 | 11 | 10 | 11 | 9 | 15 | 62
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 5 | 1 | 1 | 6 | 5 | 18
  Not Hispanic or Latino | 25 | 20 | 24 | 25 | 20 | 22 | 136
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1 | 0 | 0 | 2
  Black or African American | 2 | 1 | 1 | 3 | 2 | 0 | 9
  White | 22 | 23 | 22 | 21 | 23 | 27 | 138
  More than one race | 0 | 0 | 2 | 1 | 1 | 0 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 25.8 (2.88) | 27.2 (4.01) | 27.2 (3.55) | 25.9 (3.38) | 26.8 (3.39) | 25.9 (3.34) | 26.5 (3.42)
Baseline Average HbA1c Values [Least Squares Mean (Standard Deviation); unit: Percentage] | 7.54 (0.159) | 7.42 (0.159) | 7.58 (0.159) | 8.05 (0.153) | 7.94 (0.358) | 7.74 (0.150) | 7.71 (0.190)
Baseline Average Daily Total Insulin Use Values [Least Squares Mean (Standard Deviation); unit: Units/day] | 45.99 (3.194) | 44.21 (3.194) | 47.51 (3.194) | 42.60 (3.299) | 47.06 (3.365) | 50.03 (3.238) | 46.23 (3.247)
Time Since Type 1 Diabetes Diagnosis [Mean (Standard Deviation); unit: years] | 23.7 (10.0) | 25.1 (12.7) | 30 (13.1) | 21.7 (11.8) | 19.6 (11.7) | 25.4 (14.4) | 24.25 (12.3)

OUTCOME MEASURES:

1. Primary Outcome: Change in Average Daily Total Insulin Use
Description: Change from Baseline in average daily total insulin use at Week 12
Time Frame: Baseline and 12 weeks
Measure: Least Squares Mean (Standard Error); unit: Units/day
Groups:
- Part A - 35 mg REMD-477; Part B - 35 mg REMD-477; Part B - 70 mg REMD-477: Administered as a repeated subcutaneous (SC) doses in subjects with Type 1 Diabetes
  REMD-477: Administered as repeated SC doses in subjects with Type 1 Diabetes
- Part A - 70 mg REMD-477: Administered as a repeated SC doses in subjects with Type 1 Diabetes
  REMD-477: Administered as repeated SC doses in subjects with Type 1 Diabetes
Arm/Group | Part A - 35 mg REMD-477 | Part A - 70 mg REMD-477 | Part A - Matching Placebo | Part B - 35 mg REMD-477 | Part B - 70 mg REMD-477 | Part B - Matching Placebo
Number analyzed (Participants) | 21 | 22 | 15 | 21 | 20 | 22
Units/day | -6.72 (1.649) | -5.25 (1.634) | -1.37 (1.881) | -7.59 (2.142) | -6.64 (2.22) | -1.27 (2.103)

2. Secondary Outcome: Change From Baseline Difference in AUC Glucose Concentrations Following Mixed Meal Tolerance Test (MMTT) - Part A Only
Description: Difference from baseline at Week 13 in AUC glucose concentration following the Mixed Meal Tolerance Test (MMTT) after repeated doses of REMD-477.
Time Frame: Baseline and 13 weeks; AUC glucose timepoints: 10 minutes prior and just before (time ) initiating the mixed-meal ingestion and at 30, 60 and 120 minutes after the mixed meal ingestion.
Measure: Least Squares Mean (Standard Error); unit: min*mg/dL
Arm/Group | Part A - 35 mg REMD-477 | Part A - 70 mg REMD-477 | Part A - Matching Placebo
Number analyzed (Participants) | 23 | 23 | 21
min*mg/dL | -150.68 (40.472) | -115.05 (40.441) | -66.00 (43.020)

3. Secondary Outcome: Continuous Glucose Monitoring (CGM) - Change in Average Daily 24-hour Glucose Concentration at Week 12
Description: Change from baseline at Week 12 in average daily 24-h blood glucose as assessed by CGM after repeated doses of REMD-477.
Time Frame: Baseline and 12 weeks
Measure: Least Squares Mean (Standard Error); unit: mg/dL/day
Arm/Group | Part A - 35 mg REMD-477 | Part A - 70 mg REMD-477 | Part A - Matching Placebo | Part B - 35 mg REMD-477 | Part B - 70 mg REMD-477 | Part B - Matching Placebo
Number analyzed (Participants) | 21 | 21 | 18 | 9 | 8 | 12
mg/dL/day | 0.46 (2.561) | -5.71 (2.575) | 0.57 (2.736) | 2.57 (5.159) | -6.05 (5.435) | 6.08 (4.502)

4. Secondary Outcome: Seven-Point Glucose Profile - Change in Average 24-h Glucose Concentrations
Description: Change from baseline at Week 12 in the average daily 24-h blood glucose concentration as assessed by seven-point glucose profile after repeated doses of REMD-477. The 7-point blood glucose profiles includes measuring glucose via finger stick, at the following times of the day: before each meal, 2 hours after each meal, and at bedtime. The 7-point glucose profiles were obtained for 3 consecutive days before (Day 1) and for 3 consecutive days during week 12.
Time Frame: Baseline and 12 weeks
Population: Part A patients' compliance with the recordings of glucose values on paper diary were low, and greater than 50% of the data was missing.
Measure: Least Squares Mean (Standard Error); unit: mg/dL/day
Groups:
- Part A - 70 mg REMD-477; Part B - 70 mg REMD-477: Administered as a repeated subcutaneous (SC) doses in subjects with Type 1 Diabetes
  70 mg REMD-477: Administered as repeated SC doses in subjects with Type 1 Diabetes
- Part A - Matching Placebo; Part B - Matching Placebo: Administered as a repeated subcutaneous (SC) doses in subjects with Type 1 Diabetes
  Placebo Comparator: Administered as a repeated SC doses in subjects with Type 1 Diabetes
Arm/Group | Part A - 35 mg REMD-477 | Part A - 70 mg REMD-477 | Part A - Matching Placebo | Part B - 35 mg REMD-477 | Part B - 70 mg REMD-477 | Part B - Matching Placebo
Number analyzed (Participants) | 8 | 8 | 4 | 20 | 18 | 19
mg/dL/day | 11.02 (6.697) | -9.43 (6.830) | -4.09 (9.336) | -4.52 (9.027) | -3.71 (9.458) | 5.07 (9.091)

5. Secondary Outcome: Summary of the Product of Average Daily 24-h Glucose Ratio and Daily Insulin Use Ratio (Day 78 [Week 12]/Baseline)
Description: The product of the ratio of average glucose (Week 12/Baseline) and ratio of average insulin use (Week 12/Baseline).
Time Frame: Baseline and week 12
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | Part A - 35 mg REMD-477 | Part A - 70 mg REMD-477 | Part A - Matching Placebo | Part B - 35 mg REMD-477 | Part B - 70 mg REMD-477 | Part B - Matching Placebo
Number analyzed (Participants) | 17 | 17 | 12 | 13 | 12 | 15
Ratio | 0.86 (0.41) | 0.81 (0.041) | 0.98 (0.049) | 0.88 (0.082) | 0.89 (0.086) | 0.95 (0.077)

6. Secondary Outcome: Change in Hemoglobin A1c From Baseline at Week 13
Description: Change in Hemoglobin A1c from baseline at Week 13, after repeated doses of REMD-477.
Time Frame: Baseline and 13 weeks
Measure: Least Squares Mean (Standard Error); unit: Percentage
Arm/Group | Part A - 35 mg REMD-477 | Part A - 70 mg REMD-477 | Part A - Matching Placebo | Part B - 35 mg REMD-477 | Part B - 70 mg REMD-477 | Part B - Matching Placebo
Number analyzed (Participants) | 23 | 24 | 21 | 24 | 21 | 24
Percentage | -0.67 (0.104) | -0.66 (0.105) | -0.43 (0.109) | -0.64 (0.130) | -0.60 (0.134) | -0.11 (0.125)

7. Secondary Outcome: Percentage of Subjects With HbA1c Reduction of ≥ 0.4% at Week 13
Description: Proportion (percentage) of subjects who achieve HbA1c reduction of ≥ 0.4%, after repeated doses of REMD-477
Time Frame: Baseline and 13 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Part A - 35 mg REMD-477 | Part A - 70 mg REMD-477 | Part A - Matching Placebo | Part B - 35 mg REMD-477 | Part B - 70 mg REMD-477 | Part B - Matching Placebo
Number analyzed (Participants) | 24 | 24 | 21 | 24 | 22 | 26
Participants | 16 | 17 | 9 | 13 | 12 | 8

8. Secondary Outcome: Change in C-peptide Adjusted AUC Following Mixed Meal Tolerance Test (MMTT)
Description: Change from baseline at Week 13 in the C-peptide adjusted AUC following MMTT after repeated doses of REMD-477.
Time Frame: Baseline and 13 weeks; AUC C-peptide timepoints: 10 minutes prior and just before (time 0) initiating the mixed-meal ingestion and at 30, 60 and 120 minutes after the mixed meal ingestion.
Population: MMTT was completed in Part A subjects only. MMTT was removed from Part B as part of a protocol amendment, and Part B subjects did not complete the MMTT.
Measure: Least Squares Mean (Standard Error); unit: min*pmol/L
Arm/Group | Part A - 35 mg REMD-477 | Part A - 70 mg REMD-477 | Part A - Matching Placebo
Number analyzed (Participants) | 8 | 12 | 10
min*pmol/L | 27.33 (107.029) | 289.93 (87.212) | 166.99 (96.052)

9. Secondary Outcome: Change in Baseline Difference in Glucagon Adjusted AUC Following Mixed Meal Tolerance Test (MMTT) - Part A Only
Description: Change from baseline at Week 13 in glucagon adjusted AUC after MMTT challenge, after repeated doses of REMD-477.
Time Frame: Baseline and 13 weeks; AUC glucagon timepoints: 10 minutes prior and just before (time ) initiating the mixed-meal ingestion and at 30, 60 and 120 minutes after the mixed meal ingestion.
Population: MMTT was completed in Part A subjects only. Part B subjects did not complete the MMTT.
Measure: Least Squares Mean (Standard Error); unit: min*pmol/L
Arm/Group | Part A - 35 mg REMD-477 | Part A - 70 mg REMD-477 | Part A - Matching Placebo
Number analyzed (Participants) | 3 | 4 | 3
min*pmol/L | 2398.76 (1172.219) | 345.14 (1001.903) | 13.40 (1135.048)

10. Secondary Outcome: Proportion of Subjects With Positive Anti-REMD-477 Antibodies
Description: Proportion of subjects positive for anti-REMD-477 antibody formation.
Time Frame: Day 1 (pre-dose), Day 85 (Week 13) and Day 162 (Week 24)
Measure: Number; unit: participants
Groups:
- Parts A and B - 35 mg REMD-477: Administered as a repeated subcutaneous (SC) doses in subjects with Type 1 Diabetes
  35 mg REMD-477: Administered as repeated SC doses in subjects with Type 1 Diabetes
- Parts A and B - 70 mg REMD-477: Administered as a repeated SC doses in subjects with Type 1 Diabetes
  70 mg REMD-477: Administered as repeated SC doses in subjects with Type 1 Diabetes
- Parts A and B- Matching Placebo: Administered as a repeated SC doses in subjects with Type 1 Diabetes
  Placebo Comparator: Administered as a repeated SC doses in subjects with Type 1 Diabetes
Arm/Group | Parts A and B - 35 mg REMD-477 | Parts A and B - 70 mg REMD-477 | Parts A and B- Matching Placebo
Number analyzed (Participants) | 51 | 51 | 51
participants
  Day 1 (Pre-dose) | 2 | 4 | 5
  Day 85 (Week 13) | 1 | 1 | 4
  Day 162 (Week 24) | 2 | 5 | 4

11. Secondary Outcome: Summary of REMD-477 Plasma Concentrations
Description: REMD-477 serum-concentration after repeated doses of REMD-477.
Time Frame: Baseline (Day 1 pre-dose) and Weeks 2, 5, 9, 13 and 16.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part A - 35 mg REMD-477 | Part A - 70 mg REMD-477 | Part B - 35 mg REMD-477 | Part B - 70 mg REMD-477
Number analyzed (Participants) | 25 | 25 | 20 | 20
ng/mL
  Baseline (Day 1 Pre-dose) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Week 2 | 1070 (51.0) | 3600 (47.9) | 1390 (47.3) | 2780 (65.0)
  Week 5 | 4650 (33.9) | 12600 (68.7) | 4460 (54.7) | 11000 (33.3)
  Week 9 | 6290 (41.8) | 18200 (34) | 6550 (37.5) | 14600 (26.7)
  Week 13 | 6390 (45.9) | 19300 (33.0) | 7040 (40.6) | 15700 (27.8)
  Week 16 | 1430 (110.4) | 7020 (55.4) | 1370 (84) | 5070 (51.1)

12. Secondary Outcome: Change in Hemoglobin A1c at Week 13 in Subjects With Baseline HbA1c ≥7.5%
Description: Change in Hemoglobin A1c from baseline at Week 13, after repeated doses of REMD-477.
Time Frame: Baseline and 13 weeks
Measure: Least Squares Mean (Standard Error); unit: Percentage
Arm/Group | Part A - 35 mg REMD-477 | Part A - 70 mg REMD-477 | Part A - Matching Placebo | Part B - 35 mg REMD-477 | Part B - 70 mg REMD-477 | Part B - Matching Placebo
Number analyzed (Participants) | 13 | 9 | 12 | 16 | 17 | 15
Percentage | -1.02 (0.139) | -0.94 (0.167) | -0.70 (0.141) | -0.93 (0.173) | -0.54 (0.168) | -0.12 (0.182)

13. Secondary Outcome: Proportion of Subjects With Targeted Hemoglobin A1C (HbA1c) of ≤ 7.0% at Week 13
Description: Proportion (percentage) of subjects who achieve target HbA1c reduction of ≤ 7.0% at Week 13, after repeated doses of REMD-477
Time Frame: Baseline and 13 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Part A - 35 mg REMD-477 | Part A - 70 mg REMD-477 | Part A - Matching Placebo | Part B - 35 mg REMD-477 | Part B - 70 mg REMD-477 | Part B - Matching Placebo
Number analyzed (Participants) | 24 | 24 | 21 | 24 | 22 | 26
Participants | 16 | 19 | 9 | 12 | 8 | 4

14. Secondary Outcome: Continuous Glucose Monitoring (CGM) - Change in Percent Time Spent in Target Blood Glucose Range (70-180 mg/dL) at Week 12
Description: Change from baseline at Week 12 in percent time spent in target blood glucose range (70-180 mg/dL) after repeated doses of REMD-477.
Time Frame: Baseline and 12 weeks
Measure: Least Squares Mean (Standard Error); unit: Percentage of time spent in range
Arm/Group | Part A - 35 mg REMD-477 | Part A - 70 mg REMD-477 | Part A - Matching Placebo | Part B - 35 mg REMD-477 | Part B - 70 mg REMD-477 | Part B - Matching Placebo
Number analyzed (Participants) | 19 | 18 | 16 | 16 | 12 | 16
Percentage of time spent in range | 0.55 (2.675) | 7.38 (2.730) | 1.54 (2.903) | 1.13 (3.463) | 4.20 (3.888) | 1.19 (3.409)

15. Secondary Outcome: Continuous Glucose Monitoring (CGM) - Change in Percent Time Spent in Hyperglycemia (Blood Glucose Range >180 mg/dL) at Week 12
Description: Change from baseline at Week 12 in percent time spent in Hyperglycemia (Blood Glucose Range >180 mg/dL) after repeated doses of REMD-477.
Time Frame: Baseline and 12 weeks
Measure: Least Squares Mean (Standard Error); unit: Percentage of time spent in range
Arm/Group | Part A - 35 mg REMD-477 | Part A - 70 mg REMD-477 | Part A - Matching Placebo | Part B - 35 mg REMD-477 | Part B - 70 mg REMD-477 | Part B - Matching Placebo
Number analyzed (Participants) | 19 | 18 | 16 | 16 | 12 | 16
Percentage of time spent in range | 0.21 (2.766) | -7.99 (2.840) | -1.11 (3.015) | 1.74 (3.788) | -5.02 (4.242) | -0.65 (3.731)

16. Secondary Outcome: Continuous Glucose Monitoring (CGM) - Change in Percent Time Spent in Hypoglycemia (Blood Glucose Range <70 mg/dL) at Week 12
Description: Change from baseline at Week 12 in percent time spent in Hypoglycemia (Blood Glucose Range <70 mg/dL) after repeated doses of REMD-477.
Time Frame: Baseline and 12 weeks
Measure: Least Squares Mean (Standard Error); unit: Percentage of time spent in range
Arm/Group | Part A - 35 mg REMD-477 | Part A - 70 mg REMD-477 | Part A - Matching Placebo | Part B - 35 mg REMD-477 | Part B - 70 mg REMD-477 | Part B - Matching Placebo
Number analyzed (Participants) | 19 | 18 | 16 | 16 | 12 | 16
Percentage of time spent in range | -0.82 (0.773) | 0.05 (0.792) | -0.03 (0.483) | -2.85 (1.022) | 0.85 (1.150) | -0.59 (1.010)

17. Secondary Outcome: Continuous Glucose Monitoring (CGM) - Change in Percent Time Spent in Hypoglycemia (Blood Glucose Range <55 mg/dL) at Week 12
Description: Change from baseline at Week 12 in percent time spent in Hypoglycemia (Blood Glucose Range <55 mg/dL) after repeated doses of REMD-477.
Time Frame: Baseline and 12 weeks
Measure: Least Squares Mean (Standard Error); unit: Percentage of time spent in range
Arm/Group | Part A - 35 mg REMD-477 | Part A - 70 mg REMD-477 | Part A - Matching Placebo | Part B - 35 mg REMD-477 | Part B - 70 mg REMD-477 | Part B - Matching Placebo
Number analyzed (Participants) | 19 | 18 | 16 | 16 | 12 | 16
Percentage of time spent in range | -0.15 (0.452) | 0.27 (0.457) | -0.03 (0.483) | -1.31 (0.450) | .25 (0.512) | -0.67 (0.448)

ADVERSE EVENTS:
Time Frame: All adverse events observed by the Principal Investigator or reported by subjects are collected and recorded in the eCRF, and, for serious adverse events (SAEs), on the SAE Report form. These AEs will include the following: • All serious adverse events that occur after the subject has signed the informed consent form up to the End of Study (Week 24 Visit). • All non-serious adverse events that occur after treatment with investigational product up to the End of Study (Week 24 Visit).
Groups:
- Part B - Matching Placebo: Administered as a repeated subcutaneous (SC) doses in subjects with Type 1 Diabetes
  REMD-477: Administered as repeated SC doses in subjects with Type 1 Diabetes
Arm/Group | Part A - 35 mg REMD-477 | Part A - 70 mg REMD-477 | Part A - Matching Placebo | Part B - 35 mg REMD-477 | Part B - 70 mg REMD-477 | Part B - Matching Placebo
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25 | 0/25 | 0/26 | 0/26 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 2/25 | 1/26 | 1/26 | 2/27
Other Adverse Events (participants affected / at risk) | 20/25 | 18/25 | 20/25 | 14/26 | 18/26 | 9/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A - 35 mg REMD-477 (N=25) | Part A - 70 mg REMD-477 (N=25) | Part A - Matching Placebo (N=25) | Part B - 35 mg REMD-477 (N=26) | Part B - 70 mg REMD-477 (N=26) | Part B - Matching Placebo (N=27)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetic retinopathy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemic unconsciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A - 35 mg REMD-477 (N=25) | Part A - 70 mg REMD-477 (N=25) | Part A - Matching Placebo (N=25) | Part B - 35 mg REMD-477 (N=26) | Part B - 70 mg REMD-477 (N=26) | Part B - Matching Placebo (N=27)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 7 (9) | 2 (2) | 2 (3) | 6 (6) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1) | 4 (4) | 3 (3) | 3 (4) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 3 (3) | 2 (3) | 1 (1) | 2 (3)
Headache (Nervous system disorders) | 4 (5) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Aspartate aminotransferace increased (Investigations) | 3 (3) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferace increased (Investigations) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (3) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 2 (2)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (3) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2018-10-26): https://cdn.clinicaltrials.gov/large-docs/98/NCT03117998/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-12): https://cdn.clinicaltrials.gov/large-docs/98/NCT03117998/SAP_001.pdf